CLINICAL TRIAL: NCT06667362
Title: Frequency of Periodontal Disease in Head and Neck Cancer Patients After Radiation Therapy: a Cross Sectional Study
Brief Title: Frequency of Periodontal Disease in Head and Neck Cancer Patients After Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: HAM00212
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2023-01

CONDITIONS: Periodontal Diseases; Periodontitis
Keywords: periodontitis; head and neck cancer; radiotherapy
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
This prospective cross-sectional study evaluates the frequency and risk factors of periodontal disease in head and neck cancer patients who have undergone radiotherapy. 189 patients from three radiation centers in Cairo Governorate, Egypt will be included in the study. Periodontal status will be assessed according to the 2017 classification of periodontal diseases. Data will be collected through interviews, clinical examinations, and medical records. Potential risk factors, including tumor characteristics, treatment modalities, and oral health behaviors, will be analyzed. The findings aim to provide insights into the oral health challenges faced by these patients and inform better clinical management strategies.

DETAILED DESCRIPTION:
Introduction Cancer accounts for 12% of global deaths and poses a significant health challenge, with over 10 million new cases and 6 million fatalities annually worldwide [1]. Among them, head and neck neoplasia (HNN) is a major form of cancer in India, accounting for 23% of all cancers in males and 6% in females; Depending upon the sub-site of origin and the clinical extent of the disease the 5 -year survival varies from 20% to 90% [2]. The three most common modalities used in head and neck cancer treatment are surgical resection, radiotherapy and chemotherapy, either used singly or in combination. While these modalities are effective in eliminating the tumor, they also adversely affect the normal head and neck structures surrounding the tumor. Radiation therapy has cytotoxic effects on both normal cells and malignant cells. Direct damage to the oral structures (soft and hard tissue) commonly occurs from radio- and chemotherapy, and indirect damage may also occur from systemic toxicity. These oral complications may arise during and following cancer treatment and are commonly grouped into two broad categories: acute and chronic [3].

The reported acute oral complications are mucositis, xerostomia, dysphagia, dysgeusia, and opportunistic infections, and chronic complications such as trismus, irradiation caries, osteoradionecrosis, and changes in periodontal attachment. The long-term effects comprise alteration in vascularity of soft tissue and bone, salivary gland damage, reduction in cellularity of connective tissue, and risk of increased collagen synthesis which results in fibrosis [4]. Radiation treatment induces obliterative end- arteritis that results in soft tissue ischemia and fibrosis while the irradiated bone become hypo vascular and hypoxic [5]. The periodontium is sensitive to the effect of radiation at high doses. Diminished vascularity and cellularity of the periodontal ligament membrane with widening of periodontal space, thickening, rupturing, and disorientation of Sharpey s fibers have been reported [6].

The direct and indirect effect of high-dose radiotherapy (RT) on the periodontium results in greater risk of periodontal attachment loss and tooth loss and greater risk for the development of osteoradionecrosis[7]. The extensive periodontal destruction may occur in the absence of good oral hygiene. Periodontitis in patients scheduled for head and neck radiotherapy results in acute and chronic complications such as osteoradionecrosis. Maintenance of good oral hygiene in patients undergoing radiotherapy may reduce morbidity of the known oral and periodontal side effects [8].

Patient stated to receive the head and neck radiation therapy need dental consultation at the earliest possible time. Pre-irradiation treatment depends on patient prognosis, compliance, and residual dentition, in addition to fields, ports, dose and immediacy of radiotherapy. Diseases of teeth and supporting structures are a worrying finding in a patient about to undergo tumoricidal radiotherapy for a malignant condition in the maxillofacial region because oral pain and infection are common and a potentially serious sequence to radiotherapy for head and neck tumors in patients with healthy mouth. The loss of integrity of the gingival crevicular tissues, as a result of periodontitis and radiotherapy induced thinning of these tissues together with xerostomia, mucositis, altered diet, and poor oral hygiene that often follow high-dose radiotherapy to the jaws, can create oral problems that affect the quality of life, which can cause interruption to cancer therapy [9].

The periodontal blood vessels are affected by radiation leading to widening of periodontal ligament space and destruction of bony trabeculae which may result in increased risk of periodontal disease and altered healing with diminished capacity for bone remodeling and repair [10]. Llory et al., showed a radiation-induced downshift of periopathogens [11]. Markitziu et al. [12] and Leung et al. [13] reported that due to radiation induced hypo-salivation and a concomitant increase in plaque accumulation and shift in oral micro flora the risk of periodontal infection is also increased. Shwarze et al., found a greater number of shallow periodontal pockets in radiated patients [14]. The reduced probing pocket depth does not indicate the histological pocket depth since the probe generally penetrates coronal level of junctional epithelium due to inflammation of underlying connective tissue or may be due to disparity between probing technique, probing force, or angle of insertion of the probe [8].

Studies by Epstein et al., [15] showed that direct and indirect effects of high dose of radiotherapy on periodontium resulted in increased attachment loss [7]. Marx et al. in 1987 reported that generally increasing the doses of irradiation above 7000 rads carries the risk and severity of osteoradionecrosis [9] Marciani et al, reported that dosage can indicate potential irradiation injury [12]. Smaller irradiation doses administered at higher dose rates may be more injurious than higher doses dispensed at lower dose rates. Marques et al. in 2004 stated that radiotherapy can add to a greater or lesser degree to progression of attachment loss [16].

There is an increased gingival recession observed after radiotherapy which may be due to changes in vascularity and cellularity of periodontal ligament and hypo vascular, hypocellular, and hypoxic changes in alveolar bone. In the absence of good oral hygiene rampant periodontal destruction may occur. The gingival recession associated with radiotherapy is mainly due to reduction in gingival blood flow and alteration in immune response. The gingival recession represents loss of attachment, which is an indicator of disease progression. The gingival recession may lead to sensitivity, dental caries, and difficulty in maintenance of oral hygiene.[8] (paragraphs from new articles about effect of radiotherapy on periodontium) To our knowledge, there are no existing studies that assess the prevalence of periodontitis in head and neck cancer patients who have undergone radiotherapy. Considering the potential adverse effects of radiotherapy on oral health, we hypothesize that these patients may have a higher prevalence of periodontitis compared to the general population.

This study aimed to evaluate the frequency of periodontal disease based on the recent classification in H&N cancer patients who have received radiotherapy as well as identifying any associated risk factors for periodontal disease in those patients. The goal is to provide valuable insights into the oral health challenges faced by these patients and to inform better clinical management strategies.

Subjects and Methods

Sample size calculation:

A power analysis was designed to have adequate power to apply a statistical test of the research question regarding the prevalence of periodontitis in a sample of head and neck patients of Egyptian population. By adopting a confidence interval of (95%), a margin of error of (5%) with finite population correction and by using a prevalence of periodontitis in end-stage renal disease on hemodialysis in a sample of Egyptian population based on the results of a previous study [17]. The predicted sample size (n) was found to be (189) cases. Sample size calculation was performed using Epi info for windows version 7.2 [18].

Aim of the study:

This study aimed to evaluate the frequency of periodontal status among H&N cancer patients after radiation therapy in a sample of the Egyptian population, as well as to assess the associated risk factors.

Study design:

This prospective cross-sectional study will be conducted on 189 patients at three radiation centers in Cairo Governorate, Egypt by using direct interview, dental and periodontal examination of H&N cancer patients, in addition to using medical records for medical data collections. The design followed the Declaration of Helsinki guidelines.

The proposal will be reviewed and approved by Ahmed Maher Hospital research ethics committee. Individual patient's data will be kept confidential. The procedure will be fully explained to the patients and all the recruited patients will sign an informed consent.

Patient selection:

Patients recruitment:

Inclusion criteria: older than 18 years, of either gender, with at least six teeth in the oral cavity, and undergoing radiotherapy to the head and neck region with or without chemotherapy from (6-7 weeks). Patients of head-and-neck malignancy (squamous cell carcinoma of tongue, squamous cell carcinoma of buccal mucosa, squamous cell carcinoma of hard palate, squamous cell carcinoma of soft palate, and squamous cell carcinoma base of tongue) undergoing RT with or without chemotherapy. In all patients, both the mandible and maxilla were involved in the irradiation field.

Exclusion criteria were patients of H&N malignancy with major surgical intervention (major hard tissue resection), patients with psychiatric disorders, distant metastatic disease, bone related disorders, active untreated infection, palliative care, pregnancy, and smokers, as known that smoking is an important risk factor for periodontal disease [19] to minimize the confounders in our studied sample.

Questionnaire data:

Data will be collected by a personal interview made by the principal investigator (FA) in all patients. Patients will be asked about sex, date of birth age, systemic diseases, intake of medication, date of their last dental appointment, use of removable prosthesis, and oral hygiene habits. Information about oral hygiene habits included teeth brushing with yes or no, and how many times a day they brushed their teeth per day, if they were using a mouthwash or not.

Hospital medical records:

Cancer-related information will be collected using the hospital medical records. It included information about the tumor location, tumor-node-metastasis (TNM) staging, histologic subtype, tumor grade differentiation, type of treatment, the existence of a previously treated cancer, number of radiotherapy sessions, their total body mass index (BMI).

The sixth edition of the TNM staging system for head and neck cancers will be used to classify the tumor size (T), lymph node status (N), and metastatic status (M) [20]. Tumor grade will be classified as moderately differentiated, poorly differentiated, or undifferentiated.

Intra-observer reliability:

To assess the reliability of periodontal parameters such as pocket depth (PD) and clinical attachment loss (CAL) in the present study, a pilot study will be conducted on 10 randomly selected patients before conducting the study. The PD and CAL will be assessed before and after 24 h by the same observer in random order and analyzed by intraclass correlation (ICC) analysis.

Clinical periodontal examination:

To reduce the individual variability, all the clinical measurements will be recorded by a single calibrated investigator throughout the study (FA), in addition to radiological examination for all the participants to determine the periodontal status and periodontitis stage according to the new classification of periodontal and peri-implant diseases (2017) as: Periodontally healthy individuals are those who don't have a loss of clinical attachment (due to periodontal disease), pocket depth less than or equal to three mm, and the scores of bleeding on probing in the whole mouth less than ten percent; gingivitis patients are those with no loss of clinical attachment (due to periodontal disease), pocket depth less than or equal to three mm, and the scores of bleeding on probing in the whole mouth is more than ten percent [21].

Patients with periodontitis had at least two non-adjacent teeth. Stage I periodontitis had 1-2 mm interdental CAL with radiographic bone loss affecting less than 15% of root length and no teeth lost due to periodontitis. Stage II periodontitis had 3-4 mm interdental CAL with radiographic bone loss affecting 15-33 % of root length and no teeth lost due to periodontitis. Stage III and IV periodontitis had ≥ 5 mm interdental CAL with radiographic bone extending to middle or apical third of the root. In stage III periodontitis, a number of teeth lost due to periodontitis ≤ 4 whereas in stage IV they are > 5 teeth [22].

To determine the plaque index of the subjects, their dental plaque thickness was evaluated by probing the mesial, distal, buccal, and palatal surfaces of all teeth using a Williams periodontal probe. The plaque index of an individual was determined by summing the values obtained for each tooth and calculating the averages. To determine the plaque index, [23] reference values were taken as a basis:

* Plaque index 0: No plaque is in the area adjacent to the gingiva.
* Plaque index 1: There is a plaque in the form of a thin film on the gingival margin.
* Plaque index 2: There is a visible plaque in the gingival pocket and gingival margin.
* Plaque index 3: There is a dense plaque in the gingival pocket and on the gingival margin.

The PI had been calculated by dividing the number of plaque-containing surfaces by the total number of available surfaces. The surfaces that did not show soft plaque accumulations at the dentogingival junction had not been included in the study.

With a periodontal probe, PD and CAL were measured on six locations of the teeth (mesio-buccal/facial, mid-buccal/facial, disto-buccal/facial, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal) excluding third molar.

Loss of clinical attachment generally is measured as the distance from the CEJ to the depth of pocket. When probing depth (distance from free gingival margin to the base of sulcus/pocket) was equal to the gingival margin (distance from free gingival margin to the CEJ) this means that there is no loss of clinical attachment and attachment epithelium is still attached to the CEJ. In other words, if during measuring the pocket depth the probe didn't pass beyond the CEJ and stopped above this point, this means no loss of clinical attachment [17].

Tooth loss due to periodontitis was addressed through history taking from the patient. Patients provided history of sound teeth with great mobility that caused discomfort and difficulty of eating and mastication.

The proportion of bleeding sites 10 second after being stimulated by a standardized manual probe with a controlled force to the bottom of the sulcus/pocket at six locations (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual) on all present teeth was assessed dichotomously as a BOP score on all present teeth.

Case definition of gingivitis according to Trombilli et al., [21] is:

Probing depth ≤3 mm BOP score ≥10%, ≤30% if localized and >30% if generalized Absence of clinical attachment loss Absence of radiographic bone loss

Other clinical parameters evaluation:

The Clinical Oral Dryness Score (CODS) [24, 25, 26]:

1. Mirror sticks to buccal mucosa.
2. Mirror sticks to tongue.
3. Frothy saliva.
4. No saliva pool in floor of mouth.
5. Tongue shows loss of papillae.
6. Altered/smooth gingival architecture.
7. Glassy appearance of other oral mucosa, especially palate.
8. Tongue lobulated/fissured.
9. Active or recent (2 teeth).
10. Debris on palate (excluding under dentures). A total CODS was calculated by adding the scores from the ten features. Increased severe oral dryness is indicated by a high overall score [24].

Salivary flow rate:

Samples from patients (a day of dialysis visit) were collected between 8:00 AM and 11:00 AM to minimize effects of the diurnal variability in salivary composition. Samples were collected before meals, and talking were prohibited during the time of collection. Unstimulated whole saliva was collected for 5 min by spitting method. The collection was timed, so that flow rate (mL/min) could be measured [27]. The normal unstimulated salivary flow rate is approximately 0.3-0.4 mL/min. A diagnosis of hyposalivation is made when the unstimulated salivary flow rate is ≤0.1 mL/min [28].

The clinical assessment of oral mucositis (OM) will be carried out using the World Health Organization Oral Toxicity Scale Grading of Oral Mucositis [29]:

Grade 0: No change or erythema without pain. Grade 1: Painful areas of erythema, no ulcers. Grade 2: Areas of erythema, some painful ulcers present. Grade 3: Erythema present on most of mucosal surfaces; many painful ulcers present.

Grade 4: Erythema present on most of mucosal surfaces; extensive painful ulcers present.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age Any gender At least six remaining teeth Undergoing head and neck radiotherapy with or without chemotherapy for 6-7 weeks Head and neck malignancy including squamous cell carcinoma of the tongue, buccal mucosa, hard palate, soft palate, and base of tongue.

Both mandible and maxilla included in the radiation field

Exclusion Criteria:

* Major surgical intervention (major hard tissue resection) Psychiatric disorders Distant metastatic disease Bone-related disorders Active untreated infection Palliative care Pregnancy Smokers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include 189 participants recruited from three radiation centers in Cairo Governorate, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Loss (CAL) | Measured once during the study.
  The distance from the cementoenamel junction (CEJ) to the bottom of the periodontal pocket. It indicates the amount of attachment loss due to periodontal disease. Measured with a periodontal probe at six sites per tooth.
Probing Depth (PD) | Measured once during the study.
  The distance from the gingival margin to the bottom of the periodontal pocket. Measured with a periodontal probe at six sites per tooth.
Bleeding on Probing (BOP) | Assessed once during the study.
  Presence or absence of bleeding from the gingival sulcus 10 seconds after probing with a standardized force. Assessed at six sites per tooth.
Plaque Index (PI) | Assessed once during the study.
  A score reflecting the thickness of dental plaque present at the gingival margin. Assessed using a Williams periodontal probe and scored on a scale of 0 to 3 (0=no plaque, 3=dense plaque).
Tooth Loss due to Periodontitis | Assessed through patient history, so it covers the period prior to the study.
  Tooth Loss due to Periodontitis
Radiographic Bone Loss | Radiographs taken once during the study.
  Assessed through radiographic examination to determine the extent of bone loss around the teeth. Used in conjunction with CAL to stage periodontitis.

SECONDARY OUTCOMES:
Clinical Oral Dryness Score (CODS) | Assessed once during the study.
  A score based on ten clinical features related to oral dryness (e.g., mirror sticking to mucosa, tongue appearance, saliva characteristics). Higher scores indicate more severe dryness.
Unstimulated Salivary Flow Rate | Saliva collected once during the study, between 8:00 AM and 11:00 AM.
  The amount of saliva produced in milliliters per minute without any stimulation. Measured by collecting whole saliva for 5 minutes.
Oral Mucositis (OM) | Assessed once during the study
  Assessed using the World Health Organization Oral Toxicity Scale, which grades the severity of oral mucositis from 0 to 4 based on the presence and extent of erythema and ulcers.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher teaching Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Ethical concerns: Sharing IPD could compromise participant privacy or confidentiality, especially if the data contains sensitive information.
  Legal restrictions: There might be legal or regulatory restrictions on sharing IPD, such as data protection laws (e.g., GDPR).

REFERENCES:
- [Background] 1. Petersen PE: Oral cancer prevention and control--the approach of the World Health Organization. Oral Oncol 2009, 45(4-5):454-460 10.1016/j.oraloncology.2008.05.023. 2. Mehrotra R, Singh M, Gupta RK, Singh M, Kapoor AK: Trends of prevalence and pathological spectrum of head and neck cancers in North India. Indian Journal of Cancer 2005, 42(2). 3. Hancock PJ, Epstein JB, Sadler GR: Oral and dental management related to radiation therapy for head and neck cancer. J Can Dent Assoc 2003, 69(9):585-590. 4. Dreizen S, Daly TE, Drane JB, Brown LR: Oral complications of cancer radiotherapy. Postgrad Med 1977, 61(2):85-92 10.1080/00325481.1977.11712115. 5. Marx RE: Osteoradionecrosis: a new concept of its pathophysiology. J Oral Maxillofac Surg 1983, 41(5):283-288 10.1016/0278-2391(83)90294-x. 6. Silverman Jr S, Chierici G: Radiation Therapy of Oral Carcinoma I. Effects on Oral Tissues and Management of the Periodontium. The Journal of Periodontology 1965, 36(6):478-484 https://doi.org/10.1902/jop.1965.36.6.478. 7. Yusof ZW, Bakri MM: Severe progressive periodontal destruction due to radiation tissue injury. J Periodontol 1993, 64(12):1253-1258 10.1902/jop.1993.64.12.1253. 8. Kassim N, Sirajuddin S, Biswas S, Rafiuddin S, Apine A: Iatrogenic Damage to the Periodontium Caused by Radiation and Radiotherapy. The Open Dentistry Journal 2015, 9:182-186 10.2174/1874210601509010182. 9. Marx RE, Johnson RP: Studies in the radiobiology of osteoradionecrosis and their clinical significance. Oral Surg Oral Med Oral Pathol 1987, 64(4):379-390 10.1016/0030-4220(87)90136-8. 10. Epstein JB, Corbett T, Galler C, Stevenson-Moore P: Surgical periodontal treatment in the radiotherapy-treated head and neck cancer patient. Spec Care Dentist 1994, 14(5):182-187 10.1111/j.1754-4505.1994.tb01129.x. 11. Llory H, Dammron A, Gioanni M, Frank RM: Some population changes in oral anaerobic microorganisms, Streptococcus mutans and yeasts following irradiation of the salivry glands. Caries Res 19
- [Derived] Abou-Bakr A, Ahmed E, William H, Hassanein FEA. Frequency of periodontal disease in head and neck cancer patients after radiation therapy: a cross-sectional study. BMC Oral Health. 2025 Jul 2;25(1):1008. doi: 10.1186/s12903-025-06391-7. PMID 40604898